CLINICAL TRIAL: NCT00384345
Title: Moderate Exercise and Bright Light Treatment in Overweight Individuals
Brief Title: Exercise and Bright Light Treatment: Effects on Body Weight and Composition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Litebook Company Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-0184-BE
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2006-07

CONDITIONS: Obesity; Fatigue
Keywords: bright light treatment; exercise; body fat index; mood; sleep; fatigue
MeSH Terms: conditions — Obesity; Fatigue; Motor Activity | interventions — Ultraviolet Therapy; Exercise

INTERVENTIONS:
Device: Bright Light Therapy
Behavioral: Exercise

SUMMARY:
Bright light therapy has been used to safely and effectively treat conditions such as Seasonal Affective Disorder and to regularize sleep in patients with circadian rhythm disorder. Based on evidence of the link between bright light, serotonin, mood and carbohydrate metabolism, it has been suggested that bright light therapy can improve weight loss but the literature on the subject is sparse. Further, the literature suggests that apart from any changes in mood and carbohydrate metabolism, bright light may reduce the unpleasant side-effects of exercise and increase compliance to an exercise program.

DETAILED DESCRIPTION:
Objective: Increased physical activity is important given the concern over the growing rates of obesity. Bright light therapy has the potential to enhancing serotonin levels, impact on carbohydrate metabolism and reducing soreness and hyperthermia associated with physical activity. The aim of this study is to conduct a controlled investigation of the effects of bright light therapy and exercise on weight loss and body composition in overweight individuals.

Research Methods and Procedures: Twenty-five overweight male and female subjects will be assigned to 6 weeks of moderate exercise with or without bright light treatment. Outcome measure included changes in body mass and body composition and ratings of mood, seasonality and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Overweight subjects
* Subjects in otherwise good health
* Subjects willing to participate in a 6-week moderate exercise program
* Bedtime between 10pm and 12am; wake-up time between 6am and 8am
* Score in the median range of the Morningness/ Eveningness Questionnaire (i.e., subjects show no distinct characteristics of phase delay or phase advance)

Exclusion Criteria:

* Progressive eye disease
* History of cataracts, macular degeneration or have undergone laser corrective eye surgery in the past 30 days.
* Currently taking any medications, e.g. antibiotics, tricyclic antidepressants, that may affect photosensitivity
* History of heart disease
* History of respiratory diseases, such as asthma, emphysema
* Any severe or uncontrolled general medical condition
* Severe psychiatric disorder (as determined by psychiatrist - CMS)
* History of mania
* Grossly obese individuals with morbid obesity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24
Dates: Start 2003-09; Study Completion 2003-12

PRIMARY OUTCOMES:
The primary outcome measure will be the amount of weight loss.

SECONDARY OUTCOMES:
Secondary outcome measures will be the ratings of mood on the POMS, CES-D and SPAQ

CONTACTS AND LOCATIONS:
Overall Officials: Colin M. Shapiro, MBBCh, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada